CLINICAL TRIAL: NCT02432365
Title: Phase II Study of Weekly Paclitaxel and Cisplatin in FIGO IB2 and IIA2 Cervical Cancer Followed by Radical Hysterectomy
Brief Title: Study of Weekly Paclitaxel and Cisplatin in FIGO IB2 and IIA2 Cervical Cancer Followed by Radical Hysterectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Asian Gynecologic Oncology Group (Other); Taiwanese Gynecologic Oncology Group (Unknown)
Responsible Party: Principal Investigator, Huei-Jean Huang, MD, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGOG14-001/TGOG1008; IRB103-4781A3 (Other: Chang Gung Memorial Hospital)
Record Dates: First submitted 2015-02-10; First posted 2015-05-04 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Cervical Cancer
Keywords: Paclitaxel; Cisplatin; Cervical cancer; Radical hysterectomy; Neoadjuvant
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weekly paclitaxel and cisplatin (Experimental): 7-day cycle schedule of paclitaxel (60 mg/m2) combining with cisplatin (40 mg/m2) NAC regimen followed by radical hysterectomy and bilateral pelvic lymphadenectomy
  Interventions: Drug: paclitaxel; Drug: cisplatin; Procedure: Radical hysterectomy and bilateral pelvic lymphadenectomy

INTERVENTIONS:
Drug: paclitaxel — 7-day cycle schedule of paclitaxel (60 mg/m2)
  Other Names: Taxol
Drug: cisplatin — 7-day cycle schedule of cisplatin (40 mg/m2)
  Other Names: Kemoplat
Procedure: Radical hysterectomy and bilateral pelvic lymphadenectomy — 2 weeks after last course of neoadjuvant chemotherapy
  Other Names: RH-PLND

SUMMARY:
The purpose was to establish a quick (7-day) cycle schedule of paclitaxel (60 mg/m2) combining with cisplatin (40 mg/m2) NAC regimen could be tolerated without interfering the following surgical treatment and a favorable overall survival rate for stages IB2 and IIA2 cervical squamous cell carcinoma (SCC).

DETAILED DESCRIPTION:
This is a multi-center, open-label, Simon's 2-stage, phase II study of paclitaxel and cisplatin as neoadjuvant therapy in patients with FIGO IB2 or IIA2, squamous cell cervical carcinoma of the uterine cervix.

Primary Objectives:

• Overall survival

Secondary Objectives:

* Safety
* Progression-free survival
* Response rate
* Postoperative RT/CRT rate
* To assess Quality-of-life

An estimate of 64 evaluable patients will be enrolled in this phase II investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Women with previously untreated, histologically confirmed squamous cell carcinoma of the uterine cervix
2. HPV16-positive aged 35-70 years or HPV16-negative age <55 years
3. FIGO stage IB2 or bulky IIA, with tumor extending to the vagina within the upper one third of the vaginal wall. Bulky tumor is defined as

   1. a visible cervical tumor with the largest diameter >4 cm or (b) a cervix expanded to > 4 cm as a result of tumor infiltration by pelvic examination
   2. verified by magnetic resonance image (MRI) or 3-dimensional (D) computed tomography (CT)
4. no suspicious extrapelvic metastasis detected by MRI or 3-D CT
5. adequate marrow, liver and renal functions :hemoglobin level >= 10 g/dL, WBC count >= 3,000/mm3 or absolute neutrophil count >= 1,500/mm3, platelet count >= 100,000/mm3, serum transaminase (AST, ALT) levels <= 60 IU/mL, total serum bilirubin within normal range, serum creatinine level <= 1.5 mg/dL, and blood urea nitrogen level <=20 mg/dL
6. adequate cardiopulmonary function that tolerates the administration of study regimen and radical hysterectomy
7. Eastern Cooperative Oncology Group performance status of 0 to 1
8. had written informed consent to participate in the study
9. Appropriate organ and marrow function :

   leukocytes >=3,000/μL absolute neutrophil count >= 1,500/μL platelets >= 100,000/μL (not platelet transfusion dependent) hemoglobin >= 10 g/dL total bilirubin within normal range AST/ALT <= 2.5 X upper limit of normal range (ULN) BUN <= 20 mg/dL serum creatinine <=1.5 mg/dL or clearance > 60 mL/min
10. a negative urinary pregnancy test in a patient with child-bearing potential

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. adenocarcinoma , adenosquamous carcinoma, or small cell carcinoma
2. concurrent or history of malignant tumor(s) other than treated nonmelanoma skin cancer
3. had received surgical procedure other than cervical biopsy or cytotoxic procedure including chemotherapy, radiotherapy or therapy with biologic response modifier(s) for the cervical tumor
4. enlarged pelvic lymph node with positive aspiration cytologic or histologic study
5. participate in investigational treatment or another clinical trial for cervical cancer
6. history of allergic reaction to platinum or paclitaxel
7. uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
8. pregnant or breast feeding women

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-02; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
overall survivial | January 31, 2023 (5 years)
  The primary objective is to determinate the difference in 5-year survival rate of subjects with NAC+RH-PLND compared with standard CCRT. Based on the pilot research, the 5-year survival rate of NAC+RH-PLND is expected to be around 87.5%. Thus, a sample size of 64 subjects in NAC+RH-PLND group is required for correctly detecting a 12.5% difference between 5-year OS rate of NAC+RH-PLND group and a reference value 75% of standard CCRT in order to achieving an 80% power at a significance level 0.05.

SECONDARY OUTCOMES:
Safety (If > 6 significant G3/4 AEs occur) | January 31, 2023 (up to 5 years)
  If > 6 significant G3/4 AEs occur
Response rate (Pathological response) | Post-operative 1 month
  Pathological response will be calculated
Postoperative RT/CRT rate | Post-operative 6 months
  Postoperative RT/CCRT will be given to defined high-risk group
Quality-of-life | at completion of neoadjuvant chemotherapy
  using EORTC QLQ-C30, EORTC-QLQ-CX24
Progression-free survival | January 31, 2023 (up to 5 years)
  PFS will be evaluated using Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Jean Huang, M.D, Principal Investigator — Gynecologic oncology
Locations (5):
- Taiwan (5):
  - Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital, Chiayi City
  - Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital, Kaohsiung City
  - Department of Obstetrics and Gynecology, Chung Shan Medical University Hospital, Taichung
  - Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital, Taipei
  - Division of Gynecologic Oncology, Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital Linkou Medical Center, Taoyuan District

REFERENCES:
- See also: MedlinePlus related topics — https://medlineplus.gov/hysterectomy.html
- See also: Drug Information available for: Cisplatin — http://druginfo.nlm.nih.gov/drugportal/name/Cisplatin
- See also: Drug Information available for: Paclitaxel — https://druginfo.nlm.nih.gov/drugportal/name/Paclitaxel
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks